CLINICAL TRIAL: NCT00806988
Title: Surgical Interventions for Moderate Ischemic Mitral Regurgitation
Brief Title: Comparing the Effectiveness of a Mitral Valve Repair Procedure in Combination With Coronary Artery Bypass Grafting (CABG) Versus CABG Alone in People With Moderate Ischemic Mitral Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alan Moskowitz, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 08-1078-00003; U01HL088942 (NIH); 594 (Other: Ct Surgery Network Research Group); NCT00838786 (obsolete NCT alias)
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Mitral Valve Insufficiency; Coronary Artery Disease
Keywords: Ischemic Mitral Regurgitation; Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Coronary Artery Disease | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitral Valve Repair (Active Comparator): Participants will undergo CABG and a mitral valve repair procedure.
  Interventions: Procedure: Mitral Valve Repair; Procedure: CABG
- CABG (Active Comparator): Participants will undergo CABG.
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: Mitral Valve Repair — Surgical techniques for mitral valve repair may need to be adjusted at the discretion of the surgeon, as based on intra-operative findings that may not be previously recognized in the pre-operative evaluation. The common elements for mitral annuloplasty planned as part of this study include the following:
  1. All procedures will be performed with cardiopulmonary bypass (CPB) and with moderate hypothermia. Cannulation will be central with aortic cannulation for arterial inflow from the cardiopulmonary bypass circuit. Right atrial or bicaval (inferior and superior vena cava) drainage cannulas will be employed.
  2. The heart will be arrested with cardioplegia.
  3. A complete annular ring shall be placed unless specifically contraindicated by intra-operative findings. Additional repair of the mitral apparatus itself will be based on intra-operative findings.
  Arms: Mitral Valve Repair
Procedure: CABG — CABG will be performed using standard surgical techniques. Conduit selection and harvesting methods will not be prescribed, except that utilization of the left internal mammary artery (LIMA) is recommended when a left anterior descending (LAD) graft is indicated. The technical details of bypass grafting will not be prescribed. Complete revascularization will be performed, within the judgment of the surgical investigator.

SUMMARY:
Coronary artery bypass grafting (CABG) is a procedure that people with coronary artery disease (CAD) may undergo to increase blood flow to the heart. During a CABG procedure, people who have a leak in one of the valves in the heart-the mitral valve-may at the same time undergo a procedure that repairs the valve. This study will evaluate whether people with moderate mitral valve leakage would be better off undergoing CABG plus the mitral valve repair procedure or undergoing CABG alone.

DETAILED DESCRIPTION:
CAD occurs when the arteries that supply blood to the heart become blocked as a result of plaque buildup. In severe cases, CAD can cause chest pain, shortness of breath, and heart attack. CABG is one treatment option for people with CAD. During a CABG procedure, a healthy artery or vein from another part of the body is connected to the blocked coronary artery. Blood flow is then routed around the blockage to the heart.

After a heart attack, some people may have a leak in the mitral valve of the heart. This condition is known as ischemic mitral regurgitation (IMR) and is associated with poor health outcomes, including worsening heart failure. In people with severe mitral valve leakage, the CABG procedure and a mitral valve repair procedure are routinely performed together; however, in people with only moderate valve leakage, there is no consensus in the medical community as to whether the mitral valve repair procedure is beneficial at the time of CABG. The purpose of this study is to determine whether people with moderate mitral valve regurgitation should undergo a mitral valve repair procedure in addition to CABG or undergo CABG alone.

This study will enroll people with CAD who require a CABG procedure and have moderate mitral regurgitation. At a baseline study visit, participants will undergo a physical examination; blood collection; neurocognitive tests; and questionnaires regarding medical history, medication history, and quality of life. In the operating room, participants will be randomly assigned to undergo either CABG surgery and the mitral valve repair procedure or only CABG surgery. Blood, urine, and tissue samples may be collected from participants after the surgery; this is optional and will only be done with prior approval from participants. All participants will attend study visits at Months 6, 12, and 24. At each visit, participants will take part in a medication history review, a physical examination, an echocardiogram, a cardiopulmonary exercise test, neurocognitive tests, and quality of life surveys.

ELIGIBILITY:
Inclusion Criteria:

* Moderate mitral regurgitation in the judgment of the clinical site echocardiographer, assessed by transthoracic echocardiogram. Assessment of mitral regurgitation will be performed using an integrative method (Zoghbi W. et al. J. American Society of Echocardiography. 2003:16:777-802. see appendix). Quantitative guidelines as proposed would be: ERO between 0.2 cmsq to 0.39 cmsq. If ERO < 0.2, then the degree of mitral regurgitation will be guided by other color Doppler quantitative methods (jet area/left atrial area ratio, vena contracta, supportive criteria in an integrated fashion
* CAD that is amenable to CABG and a clinical indication for revascularization
* Age ≥ 18 years

Exclusion Criteria:

* Any evidence of structural (chordal or leaflet) mitral valve disease
* Inability to derive ERO and end-systolic volume index (ESVI) by transthoracic echocardiography
* Planned concomitant intra-operative procedures (with the exception of closure of patent foramen ovale [PFO] or atrial septal defect [ASD]or Maze procedure or left atrial appendage excision)
* Prior surgical or percutaneous mitral valve repair
* Contraindication to cardiopulmonary bypass (CPB)
* Clinical signs of cardiogenic shock at the time of surgery
* Treatment with chronic intravenous inotropic therapy at the time of surgery
* Severe, irreversible pulmonary hypertension in the judgment of the investigator
* ST segment elevation myocardial infarction (MI) requiring intervention in the 7 days before surgery
* Congenital heart disease (except PFO or ASD)
* Evidence of cirrhosis or liver synthetic failure
* Recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair compliance with the study, in the judgment of the investigator
* Therapy with an investigational intervention at the time of screening, or planning to enroll in an additional investigational intervention study during participation in the study
* Any concurrent disease with a life expectancy of less than 2 years
* Pregnancy at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2008-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, MD, Study Chair — Christiana Care Health Services; Patrick O'Gara, MD, Study Chair — Brigham and Women's Hospital; Annetine Gelijns, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Alan Moskowitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (27):
- United States (19):
  - University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - University of Maryland, Baltimore, Maryland
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Research Institute, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Toronto Sunnybrook Health Science Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - University of Toronto, Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Quebec Heart Institute/Laval Hopital, Québec, Quebec
- Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Result] Smith PK, Puskas JD, Ascheim DD, Voisine P, Gelijns AC, Moskowitz AJ, Hung JW, Parides MK, Ailawadi G, Perrault LP, Acker MA, Argenziano M, Thourani V, Gammie JS, Miller MA, Page P, Overbey JR, Bagiella E, Dagenais F, Blackstone EH, Kron IL, Goldstein DJ, Rose EA, Moquete EG, Jeffries N, Gardner TJ, O'Gara PT, Alexander JH, Michler RE; Cardiothoracic Surgical Trials Network Investigators. Surgical treatment of moderate ischemic mitral regurgitation. N Engl J Med. 2014 Dec 4;371(23):2178-88. doi: 10.1056/NEJMoa1410490. Epub 2014 Nov 18. PMID 25405390
- [Derived] Bertrand PB, Overbey JR, Zeng X, Levine RA, Ailawadi G, Acker MA, Smith PK, Thourani VH, Bagiella E, Miller MA, Gupta L, Mack MJ, Gillinov AM, Giustino G, Moskowitz AJ, Gelijns AC, Bowdish ME, O'Gara PT, Gammie JS, Hung J; Cardiothoracic Surgical Trials Network (CTSN). Progression of Tricuspid Regurgitation After Surgery for Ischemic Mitral Regurgitation. J Am Coll Cardiol. 2021 Feb 16;77(6):713-724. doi: 10.1016/j.jacc.2020.11.066. PMID 33573741
- [Derived] Capoulade R, Zeng X, Overbey JR, Ailawadi G, Alexander JH, Ascheim D, Bowdish M, Gelijns AC, Grayburn P, Kron IL, Levine RA, Mack MJ, Melnitchouk S, Michler RE, Mullen JC, O'Gara P, Parides MK, Smith P, Voisine P, Hung J; Cardiothoracic Surgical Trials Network (CTSN) Investigators. Impact of Left Ventricular to Mitral Valve Ring Mismatch on Recurrent Ischemic Mitral Regurgitation After Ring Annuloplasty. Circulation. 2016 Oct 25;134(17):1247-1256. doi: 10.1161/CIRCULATIONAHA.115.021014. PMID 27777294
- [Derived] Michler RE, Smith PK, Parides MK, Ailawadi G, Thourani V, Moskowitz AJ, Acker MA, Hung JW, Chang HL, Perrault LP, Gillinov AM, Argenziano M, Bagiella E, Overbey JR, Moquete EG, Gupta LN, Miller MA, Taddei-Peters WC, Jeffries N, Weisel RD, Rose EA, Gammie JS, DeRose JJ Jr, Puskas JD, Dagenais F, Burks SG, El-Hamamsy I, Milano CA, Atluri P, Voisine P, O'Gara PT, Gelijns AC; CTSN. Two-Year Outcomes of Surgical Treatment of Moderate Ischemic Mitral Regurgitation. N Engl J Med. 2016 May 19;374(20):1932-41. doi: 10.1056/NEJMoa1602003. Epub 2016 Apr 3. PMID 27040451
- See also: Click here for the Cardiothoracic Surgical Trials Network Web site. — http://www.ctsurgerynet.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mitral Valve Repair: Participants will undergo CABG and a mitral valve repair procedure.
  Mitral Valve Repair: Surgical techniques for mitral valve repair may need to be adjusted at the discretion of the surgeon, as based on intra-operative findings that may not be previously recognized in the pre-operative evaluation. The common elements for mitral annuloplasty planned as part of this study include the following:
  1. All procedures will be performed with cardiopulmonary bypass (CPB) and with moderate hypothermia. Cannulation will be central with aortic cannulation for arterial inflow from the cardiopulmonary bypass circuit. Right atrial or bicaval (inferior and superior vena cava) drainage cannulas will be employed.
  2. The heart will be arrested with cardioplegia.
  3. A complete annular ring shall be placed unless specifically contraindicated by intra-operative findings. Additional repair of the mitral apparatus itself will be based on intra-operative findings.
  CABG: CABG will be performed using
Period: Overall Study
Arm/Group | Mitral Valve Repair | CABG
Started | 150 | 151
Completed | 123 | 108
Not Completed | 27 | 43
Not completed — Death | 15 | 16
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Lost to Follow-up | 4 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitral Valve Repair | CABG | Total
Number analyzed (Participants) | 150 | 151 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.6) | 65.2 (11.3) | 64.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 52 | 96
  Male | 106 | 99 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 138 | 137 | 275
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 21 | 50
  White | 115 | 122 | 237
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 35 | 36 | 71
  United States | 114 | 114 | 228
  Denmark | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Degree of Left Ventricular Remodeling, as Assessed by Left Ventricular End Systolic Volume Index (LVESVI)
Time Frame: Measured at Month 12
Measure: Mean (Standard Deviation); unit: ml per square meter
Arm/Group | Mitral Valve Repair | CABG
Number analyzed (Participants) | 150 | 151
ml per square meter | 49.6 (31.5) | 46.1 (22.4)
Statistical Analysis 1: Comparison: Mitral Valve Repair vs CABG; The primary null hypothesis was that there would be no significant between-group difference in the LVESVI at 12 months; Test type: Other — An intention-to-treat analysis using a two-tailed Wilcoxon rank-sum test, at a 0.05 alpha level was used. This analysis accommodated missing LVESVI outcomes owing to death by assigning deceased patients the worst ranks in order according to the time of death. In the case of data that were missing for reasons other than death, we used multiple imputation to calculate the 12-month LVESVI on the assumption that the data were missing at random; p = 0.61, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Major Adverse Cardiac Event, Including Death, Stroke, Worsening Heart Failure (+1 New York Heart Association [NYHA] Class), Congestive Heart Failure Hospitalization, or Mitral Valve Re-intervention
Time Frame: Measured at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Repair | CABG
Number analyzed (Participants) | 150 | 151
Participants | 46 | 48
Statistical Analysis 1: Comparison: Mitral Valve Repair vs CABG; Test type: Other; p = 0.83, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Mitral Valve Repair | CABG
All-Cause Mortality (participants affected / at risk) | 15/150 | 16/151
Serious Adverse Events (participants affected / at risk) | 88/150 | 79/151
Other Adverse Events (participants affected / at risk) | 44/150 | 37/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitral Valve Repair (N=150) | CABG (N=151)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 5 (6)
Arrhythmias - Sustained ventricular arrhythmia (Cardiac disorders) | 4 (4) | 5 (5)
Arrhythmias - Sustained supraventricular arrhythmia (Cardiac disorders) | 22 (24) | 11 (11)
Pericardial Fluid Collection (Cardiac disorders) | 2 (2) | 1 (1)
Hepatic Dysfunction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Major Infection - Localized (Infections and infestations) | 18 (25) | 15 (22)
Major Infection - Endocarditis (Cardiac disorders) | 2 (2) | 1 (1)
Major Infection - Sepsis (Infections and infestations) | 8 (9) | 6 (7)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction - Peri-CABG MI (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction - Peri-Percutaneous Intervention MI (Cardiac disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - TIA (Nervous system disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - CVA-Ischemic (Nervous system disorders) | 6 (6) | 2 (2)
Neurological Dysfunction - CVA-Hemorrhagic (Nervous system disorders) | 1 (1) | 0 (0)
Neurological Dysfunction - Toxic Metabolic Encephalopathy (Nervous system disorders) | 3 (3) | 0 (0)
Neurological Dysfunction - Other (Nervous system disorders) | 4 (4) | 1 (1)
Renal dysfunction (no dialysis) (Renal and urinary disorders) | 7 (7) | 2 (2)
Renal failure (dialysis) (Renal and urinary disorders) | 5 (6) | 6 (7)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (9)
Heart Failure (Cardiac disorders) | 26 (40) | 26 (39)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 0 (0) | 2 (2)
Venous Thromboembolism Event (Vascular disorders) | 4 (4) | 3 (3)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 8 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
2 Degree AV Block Type 1 (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Aortic Aneurysm with claudication (Vascular disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute vision loss, non-neurological (Eye disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Annuloplasty ring dehiscence (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bradyarrhythmia requiring pacemaker (Cardiac disorders) | 5 (5) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia requiring pacemaker (Cardiac disorders) | 0 (0) | 1 (1)
Broken Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 2 (2)
Carotid Disease (Cardiac disorders) | 2 (2) | 1 (1)
Chest Pain/ACS (Cardiac disorders) | 3 (3) | 10 (15)
Chest Pain/ACS/PCI (Cardiac disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Coagulopathy/HIT (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Coagulopathy/HIT (-) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Contrast induced nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Depression and anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic Foot Ulcer (Vascular disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Epistaxis (Vascular disorders) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GI Bleed/GI Issue (Gastrointestinal disorders) | 7 (7) | 6 (6)
Gangrenous Toe (Vascular disorders) | 0 (0) | 1 (1)
Heart Transplant (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypoxia and respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ICD Implant (Cardiac disorders) | 2 (2) | 0 (0)
Ischemic Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischemic Left hand (Vascular disorders) | 1 (1) | 0 (0)
LV apical cannula clot (Cardiac disorders) | 1 (1) | 0 (0)
Left superficial femoral artery pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Lower extremity ischemia (Vascular disorders) | 1 (1) | 0 (0)
Malfunctioning PM (Cardiac disorders) | 1 (1) | 0 (0)
Non Sustained VT (Cardiac disorders) | 3 (3) | 0 (0)
Non-healing wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Organ Transplant (Renal and urinary disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 3 (5)
Peripheral vascular disease/BKA (Vascular disorders) | 0 (0) | 1 (1)
Pill esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Post anesthetic Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
R/O LV Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Renal Calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Small bowel obstruction/ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sternal Non-Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 3 (3) | 1 (1)
Torn aorta (Vascular disorders) | 1 (1) | 0 (0)
Hemostasis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrectomy (Renal and urinary disorders) | 1 (1) | 0 (0)
Right Axillary hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ruptured appendix (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitral Valve Repair (N=150) | CABG (N=151)
Arrhythmias - Sustained supraventricular arrhythmia (Cardiac disorders) | 24 (25) | 18 (18)
Hepatic Dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Major Infection - Localized (Infections and infestations) | 13 (19) | 9 (11)
Myocardial infarction - Peri-CABG MI (Cardiac disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - Toxic Metabolic Encephalopathy (Nervous system disorders) | 4 (4) | 0 (0)
Neurological Dysfunction - Other* (Nervous system disorders) | 2 (2) | 1 (1)
Renal dysfunction (no dialysis) (Renal and urinary disorders) | 4 (4) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Venous Thromboembolism Event (Vascular disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI Bleed/GI Issue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemetemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pressure ulcers (Vascular disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - TIA (Vascular disorders) | 1 (1) | 0 (0)
Bradyarrhythmia requiring pacemaker (Cardiac disorders) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-healing wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No